CLINICAL TRIAL: NCT01172600
Title: Effect of Nitrous Oxide in Treating Neuropathic Pain: A Pilot Study in Chronic Low Back Pain Patients
Brief Title: Effect of Nitrous Oxide in Treating Neuropathic Pain: A Study in Chronic Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Alparslan Turan, Alparslan Turan, M.D., The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10-446
Record Dates: First submitted 2010-07-27; First posted 2010-07-30 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Low Back Pain; Radiating Pain
Keywords: radiating back pain; epidural block; steroid; recurrent low back pain; Lumbar Epidural Steroid Block with 3 injections
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Entonox; Nitrous Oxide; Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Entonox (Active Comparator): Patients will receive inhaled Entonox along with the interventional block they are scheduled.
  Interventions: Other: Entonox
- Oxygen (Placebo Comparator): Patients will receive inhaled oxygen along with the interventional block they are scheduled.
  Interventions: Other: Oxygen

INTERVENTIONS:
Other: Entonox — Those randomized to Entonox will inhale the gas through a mouthpiece throughout the procedure and also continue to receive it for a total of 4 hours in the recovery.
  Other Names: Nitrous Oxide
  Arms: Entonox
Other: Oxygen — Those randomized to oxygen will inhale it through a mouthpiece throughout the procedure and also continue to receive it for a total of 4 hours in the recovery.
  Arms: Oxygen

SUMMARY:
Epidural injection will be completed under fluoroscopy and all patients will receive 1-4 mg of Midazolam for relaxation before procedure and, if needed, 50-100 mcg of Fentanyl intravenous (IV). Radiopaque contrast (Omnipaque 300), for confirming the epidural position of the needle, steroids and local anesthetic agents will be used according to the physician performing the block and will not be controlled by the study. Patients will be randomly assigned to receive either inhaled Entonox along with the interventional block they are scheduled for or oxygen. They will be blinded about the treatment they are receiving. Those randomized to Entonox will inhale the gas through a mouthpiece throughout the procedure and also continue to receive it for a total of 4 hours in the recovery. Those randomized to the oxygen group will receive oxygen through a similar mouthpiece for the entire duration of the procedure and recovery for 4 hours. Following completion of procedure the patient will be transferred to recovery and monitored for 3-5 hours then discharged home with instructions. Possible side effects will be monitored and recorded, pain score of patient will be recorded before discharge. All the patients will receive standard instructions regarding physical back exercises. This will be repeated for every procedure up to maximum of three blocks.

The patients will be followed during each block and over a period of 1, 3, 6 and 12 months and on each follow-up visit will complete computerized set of questionnaires as they did before the procedure. The patients charts will be then reviewed for one year after the initial procedure to determine if further epidural steroid injections or surgery for the presenting problem were required. It is anticipated that the appropriate number of patients will be enrolled within six months of study initiation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old at time of the first procedure
* Male or female
* History of chronic low back pain for longer than 6 months due to radiculopathy, symptomatic spinal canal stenosis, disc prolapse, postlaminectomy syndrome
* magnetic resonance imaging or electromyographic evidence of nerve root damage
* Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) score of >12
* No or minimal evidence of facet joint pathology

Exclusion Criteria:

* Known contraindications for epidural injection
* Patients with ongoing workers' compensation claims
* unstable or heavy opioid use (400 mg of morphine equivalents daily),
* psychiatric disorders
* medical illness, including conditions that could interfere with the interpretation of the outcome assessments
* pregnant or lactating women
* Current or recent drug abuse (within past 6 months).
* Patient refuses regional analgesia.
* Alcohol or drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Entonox | Oxygen
Started | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entonox | Oxygen | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (20) | 73 (16) | 71 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 22 | 18 | 40
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 27 | 27 | 54
  African American | 12 | 12 | 24
Body mass index [Median (Inter-Quartile Range); unit: kg/m2] | 30 [27 to 35] | 28 [25 to 34] | 30 [26 to 34]
American Society of Anesthesiologists physical status [Number; unit: participants]
  I: A normal healthy patient | 9 | 7 | 16
  II: A patient with mild systemic disease | 30 | 27 | 57
  III: A patient with severe systemic disease | 0 | 5 | 5
Smoking status [Number; unit: participants]
  Current Smoker | 10 | 9 | 19
  Previously quit | 15 | 12 | 27
  Never smoked | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in VAS Pain Score From Baseline to 3 Month Follow-up
Description: 10-cm-long Visual Analog Scale (VAS) pain score, ranges from 0 (no pain) to 10 (worst pain imaginable). It was measured before 1st 2nd and 3rd block and at 3 month follow-up.
  The primary outcome was the change in VAS pain score from baseline (before 1st block) to the 3 month follow-up.
Time Frame: At baseline (before 1st block) and 3 months follow-up after last block (maximum of 3 blocks with a typical 1 month interval between blocks)
Population: For 10 patients with missing VAS at 3 month follow up: 5 patients who had 2nd or 3rd epidural block, we assigned the last VAS observation (i.e., from VAS before 2nd or 3rd block to 3 month follow-up); and for 5 patients who only had 1st epidural, we assigned the worst VAS (10) for Entonox patients and the best VAS (0) for Oxygen patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 39 | 39
units on a scale | -1.6 (3.0) | -1.2 (2.6)
Statistical Analysis 1: Comparison: Entonox vs Oxygen; Test type: Superiority or Other; p = 0.84, Regression, Linear; The analysis adjusted for VAS at baseline (before 1st block), number of epidural blocks received, and imbalanced baseline variables; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-1.43 to 1.17] — This is an intention- to-treat analysis. We assigned missing outcomes to 10 patients
Statistical Analysis 2: Comparison: Entonox vs Oxygen; Test type: Superiority or Other; p = 0.12, Regression, Linear; Mean Difference (Final Values) = -1.03, 95% CI 2-sided [-2.34 to 0.28] — This is a per-protocol analysis, using 68 patients with completed data

2. Primary Outcome: Change in VAS Pain Score From Baseline to Before 2nd Block
Description: 10-cm-long Visual Analog Scale (VAS) pain score, ranges from 0 (no pain) to 10 (worst pain imaginable). It was measured before 1st 2nd and 3rd block and at 3 month follow-up.
  The primary outcome was the change in VAS pain score from baseline (before 1st block) to before the 2nd block.
Time Frame: At baseline (before 1st block) and before the 2nd block, typically at 1 month from baseline
Population: 10 patients in the Entonox group and 11 patients in the Oxygen group did not receive the 2nd block treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 29 | 28
units on a scale | -0.6 (1.7) | -0.4 (2.1)
Statistical Analysis 1: Comparison: Entonox vs Oxygen; Test type: Superiority or Other; p = 0.63, Mixed Models Analysis; Mixed model with repeated measures, adjusting for VAS pain score at baseline, number of epidural blocks received, and imbalanced baseline variables; Mean Difference (Final Values) = -0.29, 98.3% CI 2-sided [-1.80 to 1.21] — This analysis was per-protocol, using only patients with completed data

3. Primary Outcome: Change in VAS Pain Score From Baseline to Before 3rd Block
Description: 10-cm-long Visual Analog Scale (VAS) pain score, ranges from 0 (no pain) to 10 (worst pain imaginable). It was measured before 1st 2nd and 3rd block and at 3 month follow-up.
  The primary outcome was the change in VAS pain score from baseline (before 1st block) to before the 3rd block
Time Frame: At baseline (before 1st block) and before the 3rd block, typically at 2 months from baseline
Population: 21 patients in the Entonox group and 26 patients in the Oxygen group did not receive the 2nd block treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 18 | 13
units on a scale | -2.1 (3.0) | -0.5 (2.2)
Statistical Analysis 1: Comparison: Entonox vs Oxygen; Test type: Superiority or Other; p = 0.16, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.11, 98.3% CI 2-sided [-3.05 to 0.82] — This analysis was per-protocol, using only patients with completed data

4. Secondary Outcome: Change in Oswestry Score (% of Disability) From Baseline to 2nd Block
Description: Oswestry score ranges from 0% to 100%, which measures % of disability. The outcome is change in the Oswestry score from baseline (before 1st block) to before 2nd block.
Time Frame: At baseline (before 1st block) and before the 2nd block, typically at 1 month from baseline
Population: 10 Entonox patients and 11 Oxygen patients did not receive 2nd block.
Measure: Mean (Standard Deviation); unit: absolute percentage
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 29 | 28
absolute percentage | -7 (14) | -6 (14)

5. Secondary Outcome: Change in Oswestry Score (% of Disability) From Baseline to 3rd Block
Description: Oswestry score ranges from 0% to 100%, which measures % of disability. The outcome is change in the Oswestry score from baseline (before 1st block) to before 3rd block.
Time Frame: At baseline (before 1st block) and before the 3rd block, typically at 2 months from baseline
Population: 21 Entonox patients and 26 Oxygen patients did not receive 3rd block.
Measure: Mean (Standard Deviation); unit: absolute percentage
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 18 | 13
absolute percentage | -10 (13) | -7 (18)

6. Secondary Outcome: Change in Oswestry Score (% of Disability) From Baseline to 3 Months Follow-up
Description: Oswestry score ranges from 0% to 100%, which measures % of disability. The outcome is change in the Oswestry score from baseline (before 1st block) to 3 months follow-up.
Time Frame: as for outcome 1
Population: 5 patients in each group were lost follow-up.
Measure: Mean (Standard Deviation); unit: absolute percentage
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 34 | 34
absolute percentage | -11 (19) | -6 (21)

7. Secondary Outcome: Usage of Opioids
Time Frame: 2nd block, typically at 1 month from baseline
Population: 10 Entonox patients and 11 Oxygen patients did not receive 2nd block.
Measure: Number; unit: participants
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 29 | 28
participants | 3 | 7

8. Secondary Outcome: Usage of Opioid
Time Frame: 3rd block, typically at 2 months from baseline
Population: 21 Entonox patients and 26 Oxygen patients did not receive 2nd block.
Measure: Number; unit: participants
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 18 | 13
participants | 3 | 2

9. Secondary Outcome: Usage of Opioid
Time Frame: 3 months follow-up after last block (maximum of 3 blocks with a typical 1 month interval between blocks)
Population: 5 patients in each group were lost follow up.
Measure: Number; unit: participants
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 34 | 34
participants | 6 | 9

10. Secondary Outcome: Biomarkers
Description: BIOMARKERS: IL-1β, IL-6, IL-10, 1L-17A, IFN-γ, and TNF-α
Time Frame: baseline - before 1st block
Population: Blood sample was not collected for 5 Entonox patients and 1 Oxygen patients.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 34 | 38
pg/ml
  IL-1β | 206 [88 to 372] | 140 [72 to 347]
  IL-6 | 226 [126 to 458] | 198 [118 to 579]
  IL-10 | 174 [130 to 294] | 176 [143 to 397]
  IL-17A | 146 [104 to 256] | 137 [105 to 183]
  IFN-γ | 93 [77 to 176] | 85 [73 to 182]
  TNF-α | 13 [7 to 24] | 9 [5 to 24]

11. Secondary Outcome: Biomarkers
Description: BIOMARKERS: IL-1β, IL-6, IL-10, 1L-17A, IFN-γ, and TNF-α
Time Frame: before 2nd block, typically at 1 month from baseline
Population: 10 Entonox patients and 11 Oxygen patients did not come for 2nd block. Among patients came for the 2nd block, blood sample was not collected in 9 Entonox patients and 6 Oxygen patients.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 20 | 22
pg/ml
  IL-1β | 128 [64 to 289] | 100 [57 to 728]
  IL-6 | 224 [99 to 321] | 127 [99 to 797]
  IL-10 | 142 [102 to 305] | 163 [122 to 493]
  IL-17A | 146 [114 to 285] | 128 [99 to 198]
  IFN-γ | 124 [73 to 337] | 79 [63 to 129]
  TNF-α | 10 [4 to 21] | 10 [3 to 23]

12. Secondary Outcome: Biomarkers
Description: BIOMARKERS: IL-1β, IL-6, IL-10, 1L-17A, IFN-γ, and TNF-α
Time Frame: before 3rd block, typically at 2 months from baseline
Population: 21 Entonox patients and 26 Oxygen patients did come for the 3rd block. Among the patients who came for the 3rd block, blood sample was not collected in 5 Entonox patients and 1 Oxygen patient.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 13 | 12
pg/ml
  IL-1β | 120 [64 to 231] | 113 [99 to 316]
  IL-6 | 110 [90 to 258] | 239 [142 to 432]
  IL-10 | 170 [125 to 301] | 244 [146 to 651]
  IL-17A | 153 [99 to 195] | 140 [123 to 186]
  IFN-γ | 97 [69 to 138] | 88 [73 to 120]
  TNF-α | 5 [4 to 9] | 11 [7 to 13]

13. Secondary Outcome: Biomarkers
Description: BIOMARKERS: IL-1β, IL-6, IL-10, 1L-17A, IFN-γ, and TNF-α
Time Frame: 3 months follow-up after last block (maximum of 3 blocks with a typical 1 month interval between blocks)
Population: No blood sample was planned to be collected.
Arm/Group | Entonox | Oxygen
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Entonox | Oxygen
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes